CLINICAL TRIAL: NCT01937273
Title: Prospective Analysis of the Nutritional Status of Chemo-radiotherapy Patients
Brief Title: The Nutritional Status of Chemo-radiotherapy Patients
Acronym: PANSOCRP
Status: Completed | Type: Observational
Sponsor: Charles Darwin University (Other)
Responsible Party: Sponsor
Other Study IDs: HREC2013 1973
Record Dates: First submitted 2013-08-29; First posted 2013-09-09 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition; Cancer
Keywords: Nutritional status, malnutrition, chemo-radiotherapy
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Cancer patients are one of the patient groups at highest risk for the development of malnutrition. Anti-cancer treatments, such as chemotherapy and radiotherapy, can further heighten the risk due to the nutrition-related toxicities experienced during this time.

This study aims to baseline the nutritional status of chemo-radiotherapy patients undergoing treatment at the Alan Walker Cancer Care Centre (Darwin), identify contributors to nutritional deterioration and determine if there is a difference between Indigenous and non-Indigenous patients.

DETAILED DESCRIPTION:
Background: Cancer patients are at a greater risk of malnutrition. Limited data exists on the development of malnutrition during chemo - radiotherapy, particularly in rural and remote areas of Australia. Additionally, there is no data on the nutritional status of cancer patients in the Northern Territory or areas with a high proportion of Indigenous Australians. While considering the aforementioned dearth of literature, we are conducting a study in Darwin, Northern Territory of Australia. This study aims to establish a baseline of the nutritional status of chemo - radiotherapy patients undergoing treatment at the Alan Walker Cancer Care Centre (Darwin), to identify contributing factors to nutritional deterioration, and to determine if there is a difference between Indigenous and non-Indigenous patients. This study will provide a prospective analysis of malnutrition and a clear insight of nutritional status of cancer patients. It presents the first of its kind to address the nutritional status of cancer patients in Indigenous Australians.

Methods/ design: Using the Patient Generated-Subjective Global Assessment; all eligible patients will be assessed for malnutrition and consented for participation into this study. Each participant's nutritional status will be assessed at baseline, first week of treatment, final week of treatment, and at one month post treatment. Prevalence data will be analysed using percentages. Comparative data will be analysed using chi-square tests. A linear regression analysis of the results will be undertaken. Data will be analysed using SPSS version 20 (IBM SPSS).

Discussion: Weight loss and malnutrition among cancer patient is well documented, however, results from our study might appear to be more remarkable when compared with the other published data, because of our participants demographic, assessment tool used: the Patient Generated-Subjective Global Assessment has not been validated for use in Indigenous Australian Keywords: Nutritional status, malnutrition, prospective analysis, chemo-radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over undergoing curative intent chemo-radiotherapy at AWCCC
* Able to speak basic English or have an interpreter present
* Able to provide consent

Exclusion Criteria:

* Pregnant or breast feeding women
* Non-English speaking background where interpreter not available
* Change to single modality treatment (ie change from chemo-radiotherapy to chemotherapy or radiotherapy alone) or change to treatment intent (ie change from curative intent to palliative intent)
* Violent or aggressive patients to maintain the safety of investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or over) who are being treated with curative intent chemo-radiotherapy at the Alan Walker Cancer Care Centre during the data collection period
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of malnutrition amongst chemo-radiotherapy patients | 1 year

SECONDARY OUTCOMES:
The incidence of the development of malnutrition during chemo-radiotherapy | 1 year

OTHER OUTCOMES:
Factors contributing to the development of malnutrition | 1 year
The difference between Indigenous and non-Indigenous in respect to their nutritional status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Loise Moodie, Principal Investigator — Royal Darwin Hospital
Locations (1):
- Alan Walker Cancer Care Centre, Darwin, Northern Territory, Australia